CLINICAL TRIAL: NCT01148082
Title: School Response to Families Who Have Children With Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Business decision
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: PEDSVAR0010; SU-09112009-3880 (Other: Stanford University); 17105 (Other: Stanford IRB)
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Carcinomas; Squamous Cell Carcinoma; Adenocarcinoma
Keywords: Carcinomas (including Squamous Cell and Adenocarcinoma)
MeSH Terms: conditions — Carcinoma; Carcinoma, Squamous Cell; Adenocarcinoma | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Self administered Surveys
Procedure: Interviews

SUMMARY:
The purpose of this research is to investigate school response to families who have children with cancer. It is anticipated that the results of this study will enhance the support that schools can give to the population of families who have a child with cancer. The study will involve the parents in these families, the principal and an educator in the school of the child with cancer. Measurement tools will include surveys, interviews, and other relevant educational and medical documents.

ELIGIBILITY:
Inclusion Criteria:

* Patients will not be recruited. Only parents, the school principals and the teachers will be recruited.
* Subjects will be 15 sets of parents who have had school-age children treated for cancer within the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective participants will be parents/caregivers who have had school-age children treated for cancer within the last 5 years
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-09 (Estimated); Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Evidence of support | one time
  Identify significant patterns. Documents, interview, surveys and the quantitative instrument will be analyzed with an inductive cross-case analysis. Inductive analysis means that the patterns, themes, and categories emerged out of the data rather than being imposed on them prior to data collection and analysis. A cross-case analysis means that the information will be grouped together according to answers from different people, themes, perspectives or issues. Then, a content analysis will be conducted which includes the process of identifying, coding, and categorizing the primary patterns in the data. In the final step, the data will be interpreted. Interpretation, by definition, goes beyond description. Interpretation means attaching significance to what was found offering explanations, drawing conclusions, making inferences, building linkages, attaching meaning, imposing order and dealing with rival explanations

CONTACTS AND LOCATIONS:
Overall Officials: Michael Link, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States